CLINICAL TRIAL: NCT06148623
Title: Clinical Performance Testing of Philips FAST SpO2 With Masimo Pulse Oximetry Sensors Across Skin Pigmentation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Masimo Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CIP-1088
Record Dates: First submitted 2023-11-20; First posted 2023-11-28 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Test Subject (Experimental): All subjects who are enrolled into the test group and participate in data collection have the Philips FAST SpO2 with Masimo Pulse Oximetry Sensors
  Interventions: Device: Philips FAST SpO2 with Masimo Pulse Oximetry Sensors

INTERVENTIONS:
Device: Philips FAST SpO2 with Masimo Pulse Oximetry Sensors — Noninvasive pulse oximeter

SUMMARY:
Validate the performance of Philips FAST SpO2 with Masimo Pulse Oximetry Sensors in determining functional arterial oxygen saturation (SpO2) using arterial saturation (SaO2) as a reference in the range of 70-100% in subjects of varying skin pigmentation.

ELIGIBILITY:
Inclusion Criteria (Eligible Subjects):

* Subject is 18 to 50 years of age.
* Subject weighs a minimum of 110 lbs.
* Baseline heart rate ≥ 45 bpm and ≤ 90 bpm.
* Blood Pressure: Systolic BP ≤ 140 mmHg and ≥ 90 mmHg, Diastolic BP ≤ 90 mmHg and ≥ 50 mmHg, and if systolic BP is lower than 100 mmHg and/or diastolic BP is lower than 60 mmHg, subject passes an orthostatic blood pressure test.
* Hemoglobin value ≥ 11 g/dL.
* CO value ≤ 3.0% FCOHb.
* Subject can read and communicate in English and understands the study and the risks involved.

Exclusion Criteria (Ineligible Subjects) (* = per clinician discretion):

* Subject is pregnant or breastfeeding.
* Subject has a BMI > 35.
* Subject has a history of fainting (vasovagal syncope), blacking out or losing consciousness during or after a blood draw, or has a fear of blood draws.
* Subject has open wounds, inflamed tattoos, or piercings, and/or has any visible healing wounds that a medical professional determines may place them at an increased risk for participation. *
* Subject has finger deformities, nail deformities, nail polish, and/or gel/acrylic that can interfere with study device placement. *
* Subject has known drug or alcohol abuse.
* Subject uses recreational drugs. *
* Subject experiences frequent or severe headaches and/or migraine headaches, migraine auras, altitude sickness, and/or headaches accompanied by visual changes or sensitivity to light or sound.
* Subject has experienced a concussion or head injury with loss of consciousness within the past 12 months.
* Subject has any history of a stroke, myocardial infarction (heart attack), and/or seizures.
* Subject has any chronic bleeding disorder (e.g., hemophilia).
* Subject has taken anticoagulant medication within the past 30 days (excluding nonsteroidal anti-inflammatory drugs (NSAIDs)).
* Subject has donated blood within the past 4 weeks.
* Subject has any cardiac dysrhythmia (e.g., atrial fibrillation) and has not received clearance from their physician to participate.
* Subject has a known neurological and/or psychiatric disorder (e.g., schizophrenia, bipolar disorder, Multiple Sclerosis, Huntington's disease) that interferes with the subject's level of consciousness. *
* Subject has taken opioid pain medication 24 hours before the study.
* Subject has any infectious disease (e.g., Hepatitis, HIV, Tuberculosis, Flu, Malaria, Measles). *
* Subject is taking medications known to treat any type of infectious disease.
* Subject has either signs or history of peripheral ischemia or carpal tunnel syndrome.
* Subject has had invasive surgery within the past year, including but not limited to major dental surgery, appendectomy, plastic surgery, jaw surgery, major ENT surgery, major abdominal and/or pelvic surgery, heart surgery, or thoracic surgery. *
* Subject has symptoms of congestion, head cold, or other illnesses.
* Subject has been in a severe car accident(s) or a similar type of accident(s) requiring hospitalization within the past 12 months.
* Subject has any cancer or history of cancer (not including skin cancer). *
* Subject has chronic unresolved asthma, lung disease (including COPD) and/or respiratory disease.
* Subject is allergic to lidocaine, chlorhexidine, latex, adhesives, or plastic.
* Subject has a heart condition, insulin-dependent diabetes, uncontrolled hypertension, or hypercholesterolemia.
* Subject delivered vaginally, had a pregnancy terminated, had a miscarriage with hospitalization, or had a C-section within the past 6 months.
* Subject intends on participating in any heavy lifting, repetitive movement of their wrist (including riding a motorcycle, tennis), exercise (e.g., working out, riding a bike, riding a skateboard), or any activity that will put additional stress on the wrist within 24 hours following a study that involves an arterial line.
* Difficulty inserting an intravenous line in the subject's hand or arm and/or an arterial line in the radial artery of the subject's wrist.
* Subject has any medical condition which in the judgment of the investigator and/or medical staff, renders them ineligible for participation in this study or subject is deemed ineligible by the discretion of the investigator/study staff.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2023-11-13 (Actual); Primary Completion 2025-01-14 (Actual); Study Completion 2025-01-14 (Actual)

PRIMARY OUTCOMES:
Oxygen saturation performance of Philips FAST SpO2 with Masimo pulse oximetry sensors | 1-3 hours
  Performance will be determined by calculating the average root mean square (ARMS) comparing the noninvasive oxygen saturation measurement (SpO2) to the arterial oxygen saturation (SaO2) value obtained from a reference blood sample.

SECONDARY OUTCOMES:
Difference in oxygen saturation performance between three population subgroups | 1-3 hours
  Average root mean square (ARMS) will be computed for each pigmentation subgroup for light, medium, and dark skin pigmentation and the difference between the subgroup ARMS will be calculated.

CONTACTS AND LOCATIONS:
Locations (1):
- Masimo Corporation, Irvine, California, United States